CLINICAL TRIAL: NCT04802005
Title: Effects of a Short-term Aerobic Interval Exercise Program on Cardiac Fat and Function in Women With Obesity: A Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moved to another institution
Sponsor: Southern Illinois University Edwardsville (Other)
Responsible Party: Principal Investigator, Maria Fernandez Del Valle, Principal Investigator, Southern Illinois University Edwardsville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1063
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Obesity
Keywords: Cardiac fat; Cardiac function; Aerobic interval training; Cardiac Magnetic Resonance; Vascular health
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic interval (Experimental): Aerobic interval will consist of a supervised aerobic interval training sessions 3 times/week. Duration will range between 45-50 min/session depending on the exercise energy expenditure (target expenditure ~450-500kcal/session). Each interval will have a total duration of 5 min, and it will be divided into 2 periods. The first period will consist of 3 minutes of high-intensity activity at 70-85% of predicted HRmax, and for the second period the intensity will be reduced to 60-65% of predicted HRmax for 2 minutes. The training sessions will be carried out outdoors at the trails located on campus. The activity will consist of walking and/or light jogging. The speed/incline will be changed depending on the participants' heart rate and perception using the Borg's rating of perceived exertion (RPE) as needed. The RPE for the first period range will be 13-17 (15-17 at the end of the period) and 10-12 for the second period.
  Interventions: Other: Aerobic Interval Training
- Control group (No Intervention): Participants in the control group will not participate in the training programs.

INTERVENTIONS:
Other: Aerobic Interval Training — The aerobic interval training group
  Arms: Aerobic interval

SUMMARY:
The overall goal of this project is to the study the effects of an aerobic interval training program on cardiac fat, and its relationship to cardiac function using cardiac Magnetic Resonance Imaging.

ELIGIBILITY:
Inclusion Criteria:

* females, age 18-40 years old, body mass index (BMI) ≥ 30 kg/m2 and < 39.9 kg/m2, without known metabolic and/or cardiovascular disease

Exclusion Criteria:

* known CV, metabolic or pulmonary diseases or conditions, muscular-skeletal injuries (i.e. spine, knees, hips or shoulders, taking medications that affect endocrine or cardiovascular function, hypertension, being engaged in moderate intensity exercise more than two times per week or moderate-high intensity training of any type and frequency, being pregnant, cigarette smoking, having non-removable pieces or devices incompatible with DXA and CMR assessment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Changes in Cardiac Adipose Tissue (CAT) | 2 assessment points: at baseline and week 5
  CAT will be measured using cardiac Magnetic Resonance
Changes in Cardiac Function | 2 assessment points: at baseline and week 5
  Cardiac Function will be measured using cardiac Magnetic Resonance

SECONDARY OUTCOMES:
Changes in Body Composition | 2 assessment points: at baseline and week 5
  Body composition will be measured using dual-energy x-ray absorptiometry
Changes in Cardiorespiratory Function | 2 assessment points: at baseline and week 5
  Cardiorespiratory Function will be measured on a treadmill with a metabolic cart
Changes in Muscular Strength | 2 assessment points: at baseline and week 5
  Muscular Strength will be assessed through 1 repetition maximum (1RM).
Changes in Blood Pressure | 2 assessment points: at baseline and week 5
  Blood pressure will be measured using pulse wave analysis

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez Del Valle, PhD, Principal Investigator — Southern Illinois University of Edwardsville
Locations (1):
- Southern Illinois University Edwardsville, Edwardsville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No